CLINICAL TRIAL: NCT06861257
Title: Treosulfan Therapeutic Drug Monitoring in Pediatric Hematopoietic Stem Cell Transplant Recipients
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Zecca, Head of Pediatric Oncohematology Department, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: TREO
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Hematopoietic Stem Cell Transplantation; Malignant Disorders; Non-malignant Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients with a indication for HSCT and who will will receive TREO: Pediatric patients (aged 0 to 18 years) affected by malignant or non-malignant disorders and with an indication for HSCT and who will will receive TREO as part of the pre-transplant conditioning regimen, in combination with other chemotherapy agents.

SUMMARY:
One of the major challenges to improve the outcome of hematopoietic stem cell transplantation (HSCT) is the reduction of toxicity and non-relapse mortality caused by the pre-transplant conditioning regimen, while maintaining efficacy. Treosulfan (TREO) (L-treitol-1,4-bis-methanesulfonate) is a busulfan analogue with a distinct site of alkylation that results in a more favourable toxicity profile in comparison with busulfan and total body irradiation. TREO is the prodrug of L-epoxybutane, a water-soluble bifunctional alkylating agent with remarkable myeloablative and immunosuppressive properties. The use of TREO, in combination with other chemotherapy agents, as part of the conditioning regimen for hematopoietic stem cell transplantation (HSCT) in children has progressively increased during the last decade for both malignant and non-malignant disorders. Data on TREO pharmacokinetics in the pediatric population are still scarce. To date, only a few studies, including small numbers of pediatric patients, have investigated the PK profile of TREO. These studies reported high variability of TREO pharmacokinetics, and the relationship between TREO exposure, toxicity and clinical outcome is still unresolved. Therefore, therapeutic drug monitoring with a personalized approach may be an important tool to optimize outcomes in the pediatric population. The aim of the investigators' study is to characterize TREO PK/PD profiles in children undergoing HSCT and to evaluate the relationship between TREO exposure and early toxicity and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age range 0 - 18 years.
* Life expectancy > 12 weeks.
* Diagnosis of malignant or non-malignant disorder.
* Pre-HSCT Lansky / Karnofsky score ≥ 40%.
* Indication to allogeneic or autologous HSCT with TREO as part of the pre-transplant conditioning regimen.
* Negativity of pregnancy test for female patients.
* Written informed consent signed by the parents or guardians.

Exclusion Criteria:

* Absence of written informed consent signed by the parents or guardians.
* Current clinically active infectious disease (including positive HIV serology or viral RNA).
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction <40%).
* Liver dysfunction (AST/ALT ≥ 3 times institutional upper limit normal value -ULN- or bilirubin > 3 times ULN).
* Renal dysfunction: serum creatinine > 1.5 times ULN or calculated creatinine clearance < 60 ml/min/1.73 m2
* End stage irreversible multi-system organ failure.
* Pregnant or breast feeding female patient.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 70 pediatric patients (aged 0 to 18 years) affected by malignant or non-malignant disorders and with an indication for HSCT will be enrolled at 13 transplantation sites
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of patients in therapeutic range after the first dose of TREO during the pre-transplant conditioning regimen | within 24 hours from the first dose
  proposed cumulative therapeutic target AUC 4800 mg x h /L; range 3840 -6000 mg x h /L

SECONDARY OUTCOMES:
correlation between TREO exposure and early toxicity using the NCI Common Toxicity Criteria (Toxicity score 1- 5 for each organ/system) at 100 days post HSCT | 100 days post HSCT
  treo exposure is calculated by plasma concentration AUC measurement; correlation of out-of-range AUC(0-∞) and NCI grade will be analysed using the chi-square test. Intra and inter-individual variability will be estimated with a coefficient of variation (CV%).
To evaluate the inter-individual and intra-individual variability of PK profile | day 0-3
  a PK profile will be performed by collecting plasma samples for treo plasma concentration AUC measure
To study the cumulative incidence of non-relapse mortality at 100 days post HSCT | 100 days post HSCT
correlation between TREO exposure (measured by AUC) and efficacy | 1 year post HSCT
  measured as time to engraftment and donor chimerism percentage post-HSCT

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Policlinico Sant'Orsola Malpighi, Clinica Pediatrica Oncologia Ed Ematologia Pediatrica "Lalla Seràgnoli", Bologna, bOLOGNA
  - Ospedali Civili, Presidio Ospedale Dei Bambini, Oncoematologia Pediatrica e TMO, Brescia, Brescia
  - IRCCS Istituto Giannina Gaslini, U.O.S.D. Centro Trapianto di Midollo Osseo, Genova, Genova
  - Ospedale San Raffaele, U.O. Immunoematologia Pediatrica, Milan, Milano
  - Fondazione IRCCS San Gerardo dei Tintori - Clinica Pediatrica, Monza, monza-brianza
  - Azienda Ospedaliera di Padova, Oncoematologia Pediatrica, Padua, Padova
  - Fondazione IRCCS Policlinico San Matteo, S.C. Ematologia 2 - Oncoematologia Pediatrica, Pavia, pavia
  - AOU Città della Salute e della Scienza Di Torino, SC Oncoematologia Pediatrica e Centro Trapianti, Torino, torino
  - IRCCS Materno Infantile "Burlo Garofolo", SC Oncoematologia Pediatrica e SS Trapianto Di Midollo, Trieste, Trieste
  - Ospedale Donna Bambino Azienda Ospedaliera Universitaria Integrata, U.O.C. Oncoematologia Pediatrica, Verona, VR